CLINICAL TRIAL: NCT05608798
Title: Microscopic and Spectroscopic Examination of Skin Microcirculation in Healthy Individuals Using ODI Technology
Brief Title: Healthy Volunteer Study to Assess Microcirculatory Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ODI Medical AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIV-NO-22-08-040389
Record Dates: First submitted 2022-10-19; First posted 2022-11-08 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Healthy volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Examination with the ODI-Tech medical device (Other): Diffuse reflectance spectroscopy (DRS) operating within the visible wavelength region will be used for the microvascular oxygen saturation and haematocrit measurements.
  Computer-assisted microscopy (CAM) will be used for recording frames of skin microcirculation.
  Interventions: Device: ODI-Tech medical device

INTERVENTIONS:
Device: ODI-Tech medical device — The device captures and stores frames of the movement of blood in capillaries and spectra containing information on oxygen saturation. Proprietary software is used to analyse the obtained frames and spectra to calculate microvascular parameters such as functional capillary density and microvascular oxygen saturation.
  ODI-Tech can be brought to the patient's bedside and operates non-invasively. The device parts are in contact with the patient for less than 5 minutes.

SUMMARY:
The aim of the study is to obtain microvascular data from a healthy, heterogeneous population for assessing reference values for the parameters Functional Capillary Density (FCD), heterogeneity of FCD, Microvascular Oxygen Saturation (SmvO2) and Heterogeneity of SmvO2 for healthy adults with respect to gender, age, and skin type (Fitzpatrick scale)

DETAILED DESCRIPTION:
Primary objective:

• Obtain reference data of the studied microvascular parameters in a healthy, heterogeneous population

Secondary objectives:

* Determine the reproducibility of the parameters obtained using the device produced by ODI Medical
* Confirm the safety of the device produced by ODI Medical

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Subjects without signs or symptoms of acute or chronic disease and that are not treated with regular medication (contraceptive pills/IUD and oestrogen medication for menopausal symptoms are allowed). Pregnant women can be included.

Exclusion Criteria:

* Regular smokers
* Misusers of alcohol
* Misusers of drugs
* Not intact skin or reddening in the region of interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Functional Capillary Density (FCD) | Day 1, 2 assessments, minimum 1 hour between
  Expressed as mean value
Heterogeneity of FCD | Day 1, 2 assessments, minimum 1 hour between
  FCD from each frame is recorded from four quadrants in each frame where the coefficient of variation (CoV) in each frame is calculated, as well as an average CoV based on the 20 values from the same subject and session.
Microvascular Oxygen Saturation (SmvO2) | Day 1, 2 assessments, minimum 1 hour between
  Percent
Heterogeneity of SmvO2 | Day 1, 2 assessments, minimum 1 hour between
  [coefficient of variation] within the specific assessment and patient
Tissue haematocrit (TH) | Day 1, 2 assessments, minimum 1 hour between
  Percentage
Heterogeneity of TH | Day 1, 2 assessments, minimum 1 hour between
  [coefficient of variation] within the specific assessment and patient
Visual assessment of capillary morphology | Day 1, 2 assessments, minimum 1 hour between
  dilatation, elongation, microvascular bleedings

SECONDARY OUTCOMES:
Incidence of AE/ADE/SAE/SADE/DD | Day 1
  Descriptive as number of reported, graded
Reproducibility | Day 1
  Variance of FCD, SmvO2 and its associated heterogeneity between measurements

CONTACTS AND LOCATIONS:
Overall Officials: Knut Kvernebo, PhD, MD, Study Chair — ODI Medical
Locations (1):
- ODI Medical, Oslo, Norway

REFERENCES:
- [Background] Sundheim LK, Sporastoyl AH, Wester T, Salerud G, Kvernebo K. Acute skin trauma induces hyperemia, but superficial papillary nutritive perfusion remains unchanged. Microcirculation. 2017 Oct;24(7). doi: 10.1111/micc.12389. PMID 28632939
- [Background] Fredly S, Fugelseth D, Nygaard CS, Salerud EG, Stiris T, Kvernebo K. Noninvasive assessments of oxygen delivery from the microcirculation to skin in hypothermia-treated asphyxiated newborn infants. Pediatr Res. 2016 Jun;79(6):902-6. doi: 10.1038/pr.2016.16. Epub 2016 Feb 8. PMID 26854800
- [Background] Mork C, Salerud EG, Asker CL, Kvernebo K. The prostaglandin E1 analog misoprostol reduces symptoms and microvascular arteriovenous shunting in erythromelalgia-a double-blind, crossover, placebo-compared study. J Invest Dermatol. 2004 Mar;122(3):587-93. doi: 10.1111/j.0022-202X.2004.22339.x. PMID 15086539
- [Background] Wester T, Awan ZA, Kvernebo TS, Salerud G, Kvernebo K. Skin microvascular morphology and hemodynamics during treatment with veno-arterial extra-corporeal membrane oxygenation. Clin Hemorheol Microcirc. 2014;56(2):119-31. doi: 10.3233/CH-131670. PMID 23357861
- [Background] Mork C, Kvernebo K, Asker CL, Salerud EG. Reduced skin capillary density during attacks of erythromelalgia implies arteriovenous shunting as pathogenetic mechanism. J Invest Dermatol. 2002 Oct;119(4):949-53. doi: 10.1046/j.1523-1747.2002.00218.x. PMID 12406343
- [Background] Mork C, Asker CL, Salerud EG, Kvernebo K. Microvascular arteriovenous shunting is a probable pathogenetic mechanism in erythromelalgia. J Invest Dermatol. 2000 Apr;114(4):643-6. doi: 10.1046/j.1523-1747.2000.00944.x. PMID 10733667
- [Background] Staxrud LE, Jakobsson A, Kvernebo K, Salerud EG. Spatial and temporal evaluation of locally induced skin trauma recorded with laser Doppler techniques. Microvasc Res. 1996 Jan;51(1):69-79. doi: 10.1006/mvre.1996.0008. PMID 8812758
- [Background] Bungum L, Kvernebo K, Oian P, Maltau JM. Laser doppler-recorded reactive hyperaemia in the forearm skin during the menstrual cycle. Br J Obstet Gynaecol. 1996 Jan;103(1):70-5. doi: 10.1111/j.1471-0528.1996.tb09517.x. PMID 8608101
- [Background] Fredly S, Fugelseth D, Wester T, Haggblad E, Kvernebo K. Skin microcirculation in healthy term newborn infants--assessment of morphology, perfusion and oxygenation. Clin Hemorheol Microcirc. 2015;59(4):309-22. doi: 10.3233/CH-131764. PMID 24002120
- [Background] Awan ZA, Haggblad E, Wester T, Kvernebo MS, Halvorsen PS, Kvernebo K. Diffuse reflectance spectroscopy: Systemic and microvascular oxygen saturation is linearly correlated and hypoxia leads to increased spatial heterogeneity of microvascular saturation. Microvasc Res. 2011 May;81(3):245-51. doi: 10.1016/j.mvr.2011.02.004. Epub 2011 Mar 2. PMID 21376735
- [Background] Kvernebo AK, Miyamoto T, Sporastoyl AH, Wikslund LK, Masoy SE, Drolsum L, Moe MC, Salerud G, Fukamachi K, Kvernebo K. Quantification of ocular surface microcirculation by computer assisted video microscopy and diffuse reflectance spectroscopy. Exp Eye Res. 2020 Dec;201:108312. doi: 10.1016/j.exer.2020.108312. Epub 2020 Oct 22. PMID 33157128